CLINICAL TRIAL: NCT06173596
Title: A Phase 1 Study to Evaluate the Potential Drug Interactions Between ALXN2080 and Itraconazole, Fluconazole, and Carbamazepine in Healthy Adult Participants
Brief Title: A Study to Evaluate Potential Drug Interactions Between ALXN2080 and Itraconazole, Fluconazole & Carbamazepine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D7420C00003
Record Dates: First submitted 2023-12-05; First posted 2023-12-15 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: ALXN2080; itraconazole; Fluconazole; carbamazepine
MeSH Terms: interventions — Itraconazole; Fluconazole; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): During Part 1, Period 1, participants will receive a single dose of ALXN2080 on the morning of Day 1. In Part 1, Period 2, participants will receive a dose of itraconazole orally once daily on the morning of Day 1 to Day 13. On the morning of Day 5, participants will be given a single dose of ALXN2080 co-administered with itraconazole.
  Interventions: Drug: ALXN2080; Drug: Itraconazole
- Part 2 (Optional) (Experimental): During Part 2, Period 1, participants will receive a single dose of ALXN2080 on the morning of Day 1. In Part 2, Period 2, participants will receive a single loading dose of fluconazole, followed by a dose of fluconazole qd on the morning of Day 2 to Day 10. On the morning of Day 4, participants will be given a single dose of ALXN2080 co-administered with fluconazole.
  Interventions: Drug: ALXN2080; Drug: Fluconazole (AxMP)
- Part 3 (Experimental): During Part 3, Period 1 participants will receive a single dose of ALXN2080 on the morning of Day 1. In Part 3, Period 2, participants will receive a dose of carbamazepine bid on the morning and evening of Day 1 to Day 3, followed by a dose of carbamazepine bid on the morning and evening of Day 4 to Day 6 and a dose of carbamazepine bid on the morning and evening of Day 7 to Day 23. On the morning of Day 19, participants will be given a single dose of ALXN2080 co-administered with carbamazepine.
  Interventions: Drug: ALXN2080; Drug: Carbamazepine (AxMP)

INTERVENTIONS:
Drug: ALXN2080 — Participants will receive ALXN2080 orally.
Drug: Itraconazole — Participants will receive Itraconazole orally.
  Arms: Part 1
Drug: Fluconazole (AxMP) — Participants will receive Fluconazole orally.
  Arms: Part 2 (Optional)
Drug: Carbamazepine (AxMP) — Participants will receive Carbamazepine orally.
  Arms: Part 3

SUMMARY:
The primary objectives of this study are to determine the effect of multiple doses of itraconazole on the single dose PK of ALXN2080, to determine the effect of multiple doses of fluconazole on the single dose PK of ALXN2080 (optional), and to determine the effect of multiple doses of carbamazepine on the single dose PK of ALXN2080.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs, triplicate 12-lead ECG, screening clinical laboratory profiles (hematology, clinical chemistry, coagulation, and urinalysis), as deemed by the Investigator or designee.
* Female participants of childbearing potential and male participants must follow protocol-specified contraception guidance
* BMI within the range of 18.0 to 32.0 kg/m2 (inclusive) and a minimum body weight of 50.0 kg at screening.

Exclusion Criteria:

* History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological, psychiatric or other disorders; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* History of meningococcal infection.
* History of additional risk factors for Torsades de Pointes (eg, heart failure, hypokalemia, family history of Long QT syndrome).
* History of unexplained, recurrent infection, or infection requiring treatment with systemic antibiotics within 14 days prior to Period 1 Day 1.
* History of significant multiple and/or severe allergies (hay fever is allowed unless it is active), including significant hypersensitivity reactions to commonly used antibacterial agents, including beta-lactams, penicillin, amoxicillin, aminopenicillin, fluoroquinolones (specifically including ciprofloxacin), cephalosporins, and carbapenems, which in the opinion of the Investigator would make it difficult to provide empiric antibiotic therapy or treat an active infection.
* Diseases or conditions or previous procedures known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History of malignancy within 5 years prior to screening, with the exception of nonmelanoma skin cancer or carcinoma in situ of the cervix that has been treated with no evidence of recurrence.
* Known hepatic or biliary abnormalities (including participants with Gilbert's syndrome).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ALXN2080 | Day 1 up to Day 24
Area Under the Curve From Time 0 to the Time of Last Measurable Concentration (AUC0-last) of ALXN2080 | Day 1 up to Day 24

SECONDARY OUTCOMES:
Cmax of Itraconazole | Day 4 up to Day 6
Area under the Curve for the Defined Interval Between Doses AUC(tau) of Itraconazole | Day 4 up to Day 6
Cmax of Fluconazole | Day 2 up to Day 5
AUC(tau) of Fluconazole | Day 2 up to Day 5
Cmax of Carbamazepine | Day 2 up to Day 20
AUC(tau) of Carbamazepine | Day 2 up to Day 20
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Baseline up to Day 34

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR